CLINICAL TRIAL: NCT04071886
Title: Effect of Short-Term Mindfulness-Based Training For Major Depression Disorder: An Eye-Tracking Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Lingjiang Li, President of Chinese Psychiatry Society of Chinese Medical Association, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Second Xiangya hospital EMEN
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: MDD
Keywords: eye-tracking; eye movement; mindfulness
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Training (Experimental): Participants in the Mindfulness-Based Training arm will receive 2 weeks of Mindfulness-Based Training for at least 30 minutes every day.
  Interventions: Behavioral: Mindfulness-Based Training
- Relaxation Training (Active Comparator): Participants in the Relaxation Training arm will receive 2 weeks of Relaxation Training for at least 30 minutes every day.
  Interventions: Behavioral: Relaxation Training

INTERVENTIONS:
Behavioral: Mindfulness-Based Training — Mindfulness-Based Training comprises of mindful walking, body scanning and raisin meditation exercise. Participants will receive a guided session of mindfulness meditation, and will be asked to finish at least 30 minutes of Mindfulness-Based Training every day as homework as well as keep a diary describing their experiences and reflections. An expert in mindfulness practice will offer feedback and answer any questions online.
  Arms: Mindfulness-Based Training
Behavioral: Relaxation Training — Participants will listen to a 15-minute Relaxation Training tape twice a day.
  Arms: Relaxation Training

SUMMARY:
The purpose of this study is to investigate the short-term effects of mindfulness-based training in individuals suffering from major depressive disorder (MDD) as assessed by clinical interviewing, self-report assessment, cognitive evaluation and eye-tracking task.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual (DSM-IV) diagnosis of depression
* Consent to participate in the study and to be randomized to one of two groups

Exclusion Criteria:

* Current or past substance abuse, psychotic disorder,obsessive compulsive disorder , Post-Traumatic Stress Disorder, in the past 6 months
* History of epilepsy or head trauma
* Eye disorders
* History of electroconvulsive therapy in the past 4 weeks.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Eye Movement Performance During Free-View Task at 2 Weeks | at baseline and in 2 weeks
  The first fixated location and latency (msec) of each trial, the total dwell time (msec) in each interest area (IA) during the whole trial to assess the attentional bias in the experiment.

SECONDARY OUTCOMES:
Mean Change from Baseline in the Symptoms of Major Depression as Measured by BDI-II at 2 Weeks | at baseline and in 2 weeks
  Measured by Beck Depression Inventory (BDI-II). BDI-II is a self-report questionnaire that measures the severity of depression on a scale of 0 to 63. Higher total scores indicate more severe depressive symptoms.
Mean Change from Baseline in the Symptoms of Major Depression as Measured by HAM-D at 2 Weeks | at baseline and in 2 weeks
  Measured by Hamilton Rating Scale for Depression (HAM-D). HAM-D is used by clinicians to rate the severity of depression and to evaluate recovery. HAM-D score ranges from 0 to 51, with higher scores indicating more severe depressive symptoms.
Mean Change from Baseline in State Mindfulness at 2 Weeks | at baseline and in 2 weeks
  Measured by the Five Facet Mindfulness Questionnaire (FFMQ). FFMQ measures five mindfulness skills through these subscales: Non-Reactivity to Inner Experience, Observing/Noticing, Acting With Awareness, Describing, and Non-Judging of Experience. The five subscale scores can be combined to yield a total score ranging from 0 to 195, measuring global mindfulness skills, with higher scores indicating higher level of global mindfulness skills. For FFMQ subscales, scores range from 8 to 40, except for Non-Reactivity to Experience scores, which range from 7 to 35. Higher subscale scores indicate higher level of respective mindfulness skills.
Mean Change from Baseline in Tendency to Engage in Ruminative Responses at 2 Weeks | at baseline and in 2 weeks
  Measured by the Ruminative Responses Scale of the Response Styles Questionnaire (RRS). RRS measures the tendency to ruminate. RRS score ranges from 22 to 88, with higher scores indicate a stronger tendency to engage in ruminative thoughts.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute & Faculty of Psychiatry of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No